CLINICAL TRIAL: NCT03085719
Title: Targeting PD-1 Therapy Resistance With Focused High or High and Low Dose Radiation in Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Targeting PD-1 Therapy Resistance With Focused High or High and Low Dose Radiation in SCCHN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jonathan Schoenfeld, MD, MPH, MD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-604
Record Dates: First submitted 2017-03-10; First posted 2017-03-21 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Radiation + Pembrolizumab (Experimental): * High dose radiation will be given in 3 fractions
  * Pembrolizumab administered intravenously on day one of each cycle.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation
- High Dose + Low Dose Radiation + Pembrolizumab (Experimental): * High Dose radiation will be given in 3 fractions
  * Low Dose Radiation will be given in 2 fractions
  * Pembrolizumab administered intravenously on day one of each cycle.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation

INTERVENTIONS:
Drug: Pembrolizumab — Keytruda is designed to restore the natural ability of the immune system to recognize and target cancer cells
  Other Names: Keytruda
Radiation: Radiation — Radiation is used to shrink the cancer

SUMMARY:
This research study is studying immunotherapy in combination with radiation therapy as a possible treatment for head & neck cancer that has worsened or spread to another organ or part of your body.

The immunotherapy involved in this study is: MK-3475 (pembrolizumab or KEYTRUDA).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational treatment to learn whether the treatment works in treating a specific disease. "Investigational" means that the treatment is being studied.

MK-3475 is a humanized monoclonal antibody. An antibody is a common type of protein made in the body in response to a foreign substance (particles not typically found in the body such as bacteria or viruses). Antibodies attack foreign substances and protect against infection. Antibodies can also be produced in the laboratory for use in treating patients. MK-3475 is designed to restore the natural ability of the immune system to recognize and target cancer cells.

The FDA recently granted approval to MK-3475 as a treatment for patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC). This study is testing whether using radiation in combination with MK-3475 will make this drug work better in participants that might otherwise be unlikely to benefit from this drug because they have not responded to either this same drug given without radiation or another similar drug.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma of the head and neck with evidence of metastatic disease considered incurable by local therapies. Patients without pathologic or cytologic evidence of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Patients must have evidence of radiologic or clinical disease progression during previous treatment with systemic PD-1 directed therapy, or have stable disease on prior PD-1 therapy (at least 6 doses) and/or have been deemed not to derive clinical benefit from PD-1 directed treatment.
* Patients must have least 3 measurable non-CNS based lesions that have not previously been irradiated. Palliative radiation must be potentially indicated for at least one of these lesions.
* Patients must agree to undergo a research biopsy, if tumor is accessible, at baseline (mandatory) and at the end of cycle 2 of pembrolizumab (optional). .
* Prior systemic therapy: Patients must be at least 2 weeks from prior chemotherapy, biological agents, immunotherapy or any investigational drug product, with adequate recovery of toxicity. For investigational agents, the minimum time from prior therapy is 5 half-lives if this is longer than 2 weeks in duration.
* Prior radiation therapy: Patients must be at least 2 weeks from prior radiation therapy
* Concurrent administration of other cancer specific therapy during the course of this study is not allowed.
* Only patients 18 years and older are eligible. There is no upper age limit but the patients must be able to medically tolerate the regimen. Adverse event data are currently unavailable on the use immune checkpoint blockade for participants < 18 years of age, and thus children are excluded from this study.
* ECOG performance status <=1 (see Appendix A).
* Ability to understand and the willingness to sign a written informed consent document
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
* Female and male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in section 5.7.1. Contraception is required prior to study entry and for the duration of study participation and 4 months after completion of pembrolizumab administration.

  --Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcl
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin >= 9 g/dl
  * total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN
  * AST(SGOT)/ALT(SGPT) For patients with documented liver metastases, ≤ 5 × institutional ULN
  * creatinine ≤1.5 ×within normal institutional ULN OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional ULN.
  * International normalized ratio (INR) or Prothrombin Time (PT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
  * Activated Partial Thromboplastin Time (aPTT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Laboratory tests required for eligibility must be completed within 14 days prior study entry. Baseline tumor measurements must be documented from tests within 28 days of study entry. Other non-laboratory tests must be performed within 28 days of study entry.

Exclusion Criteria:

* Metastatic disease impinging on the spinal cord or threatening spinal cord compression.
* Surgical fixation of bone lesion to be irradiated is required and indicated to provide mechanical stability.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least 2 weeks prior to trial therapy initiation, are neurologically stable, and have recovered from the acute effects of radiotherapy or surgery. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before the initiating protocol therapy. Treatment for brain metastases may include surgery, whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or previous toxicity attributed to pembrolizumab or other PD-1 directed therapy that led to drug discontinuation.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Clinically significant electrocardiogram (ECG) abnormality, including a marked Baseline prolonged QT/QTc ([QT interval/corrected QT interval], e.g., a repeated demonstration of a QTc interval >500 ms).
* Pregnant women are excluded from this study because immunotherapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with immunotherapy, breastfeeding should be discontinued if the mother is treated on this protocol.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; or if diagnosed and treated for cervical cancer in situ or basal cell or squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for interaction between immunotherapy and these medications.
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non infectious pneumonitis.
* Active, suspected or prior documented autoimmune disease that has required systemic treatment in the last 2 years with immune modifying agents (e.g. replacement therapy such as thyroxine, insulin or physiologic corticosteroids is not an exclusion criteria).
* The subject is known to be positive for HepBsAg, or HCV RNA.
* Lack of availability for follow up assessments.
* The investigator's belief that the subject is medically unfit to receive pembrolizumab and or unsuitable for any other reason.
* Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2027-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Schoenfeld, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Radiation + Pembrolizumab: * High dose radiation will be given in 3 fractions
  * Pembrolizumab administered intravenously on day one of each cycle.
  Pembrolizumab: Keytruda is designed to restore the natural ability of the immune system to recognize and target cancer cells
  Radiation: Radiation is used to shrink the cancer
- High Dose + Low Dose Radiation + Pembrolizumab: * High Dose radiation will be given in 3 fractions
  * Low Dose Radiation will be given in 2 fractions
  * Pembrolizumab administered intravenously on day one of each cycle.
  Pembrolizumab: Keytruda is designed to restore the natural ability of the immune system to recognize and target cancer cells
  Radiation: Radiation is used to shrink the cancer
Period: Overall Study
Arm/Group | High Dose Radiation + Pembrolizumab | High Dose + Low Dose Radiation + Pembrolizumab
Started | 6 | 12
Completed | 6 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The groups of 'High Dose Radiation + Pembrolizumab' and 'High Dose + Low Dose Radiation + Pembrolizumab' listed in the Participant Flow and Baseline Characteristics were the predefined groups in the study protocol; this was not a dose escalation study for pembrolizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Radiation + Pembrolizumab | High Dose + Low Dose Radiation + Pembrolizumab | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 9 | 10
Age, Continuous [Median (Full Range); unit: years] | 59 [47 to 71] | 67 [54 to 73] | 65.5 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 9 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 12 | 18
ECOG PS [Count of Participants; unit: Participants] — Participants were graded using the ECOG Performance Status (PS) Scale, which describes their ability to care for themselves and their physical ability (walking, working, etc.). An ECOG PS of 0 indicates that the participant was fully active with no restriction. An ECOG PS of 2 indicates that the participant was ambulatory and capable of all selfcare but unable to carry out any work activities.
  Participants
    0 | 0 | 2 | 2
    1 | 6 | 9 | 15
    2 | 0 | 1 | 1
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 0 | 3 | 3
  Former Smoker | 5 | 4 | 9
  Never Smoked | 1 | 5 | 6
T Stage [Count of Participants; unit: Participants] — The T Stage was determined based on the size and depth of invasion of the primary tumor (AJCC 8th Edition Staging). A higher T Stage indicates that the primary tumor is larger or exhibits a higher depth of invasion. TX means that the primary tumor could not be measured.
  Participants
    T1 | 1 | 1 | 2
    T2 | 1 | 2 | 3
    T3 | 2 | 3 | 5
    T4 | 1 | 3 | 4
    TX | 1 | 2 | 3
    Missing | 0 | 1 | 1
N Stage [Count of Participants; unit: Participants] — The N Stage was determined based on regional lymph node involvement of the tumor (AJCC 8th Edition Staging). N0 indicates no regional lymph node metastasis, while N3 indicates a higher degree of regional lymph node involvement. NX means that the regional lymph nodes could not be measured.
  Participants
    N0 | 0 | 1 | 1
    N1 | 0 | 1 | 1
    N2 | 6 | 7 | 13
    N3 | 0 | 1 | 1
    NX | 0 | 1 | 1
    Missing | 0 | 1 | 1
M Stage [Count of Participants; unit: Participants] — The M Stage describes the presence of distant metastases of the primary tumor (AJCC 8th Edition Staging). M0 classifies a tumor with no distant metastasis, and M1 classifies a tumor with evidence of distant metastasis.
  Participants
    M0 | 3 | 6 | 9
    M1 | 1 | 5 | 6
    Missing | 2 | 1 | 3
Disease Stage [Count of Participants; unit: Participants] — The Disease Stage describes the overall stage of the cancer based on the T, N, and M stages (AJCC 8th Edition Staging). A higher Disease Stage indicates that the cancer is more advanced, with Stage IV being the most advanced.
  Participants
    Stage III | 1 | 2 | 3
    Stage IV | 5 | 9 | 14
    Missing | 0 | 1 | 1
Disease Site [Count of Participants; unit: Participants]
  Oropharynx | 3 | 6 | 9
  Hypopharynx | 1 | 2 | 3
  Oral Cavity | 1 | 2 | 3
  Larynx | 1 | 1 | 2
  Other | 0 | 1 | 1
Pathology [Count of Participants; unit: Participants]
  Squamous Cell Carcinoma | 6 | 12 | 18
  Other | 0 | 0 | 0
HIV Status [Count of Participants; unit: Participants]
  Negative | 6 | 11 | 17
  Unknown | 0 | 1 | 1
HPV Status [Count of Participants; unit: Participants]
  Negative | 1 | 3 | 4
  Positive | 3 | 5 | 8
  Unknown | 2 | 4 | 6
Prior Treatment [Count of Participants; unit: Participants]
  Chemotherapy | 5 | 12 | 17
  Surgery | 4 | 5 | 9
  Radiation Therapy | 6 | 11 | 17
Prior IO Therapy Type [Count of Participants; unit: Participants]
  Nivolumab | 3 | 3 | 6
  Nivolumab/Lirilumab | 1 | 8 | 9
  Pembrolizumab | 2 | 0 | 2
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Surival
Description: The primary endpoint of this study is progression-free survival (PFS) rate at 3 months. Patients are considered progression-free at 3 months if progression is not observed at the 3-month disease assessment. PFS is defined as the time from registration to disease progression per RECIST or death, whichever occurred first.
  Progressive Disease is defined as at least a 20% increase in the sum of diameters of target lesions, which must also demonstrate an absolute increase of at least 5 mm (with reference to the smallest sum on study). The appearance of one or more new lesions is also considered progressions (RECIST guidelines version 1.1).
Time Frame: 1 year
Population: The groups of 'High Dose Radiation + Pembrolizumab' and 'High Dose + Low Dose Radiation + Pembrolizumab' listed under Primary Outcome were the predefined groups in the study protocol; this was not a dose escalation study for pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Radiation + Pembrolizumab | High Dose + Low Dose Radiation + Pembrolizumab
Number analyzed (Participants) | 6 | 12
Participants | 1 | 8

2. Secondary Outcome: Overall Survival
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Overall Response Rate
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

4. Secondary Outcome: Number of Patients With Treatment Related Adverse Events as Assessed by CTCAE v4.0
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

5. Secondary Outcome: Objective Response by Immune Related Response Criteria (irRC)
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

6. Secondary Outcome: Local Response Determined Using CT Imaging
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

7. Secondary Outcome: Clinical Benefit Rate
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: Abscopal Response Determined Using CT Imaging
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from baseline through the end of treatment (30 days after the last study intervention), for a maximum total duration of 15 months. This time period varied depending on how many total treatment cycles each patient was given.
Description: All toxicities that were definitely, probably, possibly, or not related to protocol treatment were included.
  The groups of 'High Dose Radiation + Pembrolizumab' and 'High Dose + Low Dose Radiation + Pembrolizumab' listed in Adverse Events were the predefined groups in the study protocol; this was not a dose escalation study for pembrolizumab.
Arm/Group | High Dose Radiation + Pembrolizumab | High Dose + Low Dose Radiation + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/6 | 10/12
Serious Adverse Events (participants affected / at risk) | 3/6 | 7/12
Other Adverse Events (participants affected / at risk) | 4/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Radiation + Pembrolizumab (N=6) | High Dose + Low Dose Radiation + Pembrolizumab (N=12)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral/nasal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Eye infection (Eye disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Radiation + Pembrolizumab (N=6) | High Dose + Low Dose Radiation + Pembrolizumab (N=12)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 6 (6)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Tumor site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema Face (General disorders) | 1 (1) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 4 (5)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Neck edema (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03085719/Prot_SAP_001.pdf